CLINICAL TRIAL: NCT06272292
Title: An Integrated Biomechanical Investigation of Subjects With Symptomatic FAI and Two Groups of Asymptomatic Controls: a Comparison in Dynamic Tasks
Brief Title: Biomechanical Investigation of Symptomatic FAI and Two Groups of Asymptomatic Controls
Acronym: CAM-FAI adult
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S66441
Record Dates: First submitted 2023-12-06; First posted 2024-02-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Intervention Model Description: Cross-sectional, case-control prospective clinical study
Who Masked: Participant
Masking Description: 3 study groups, based on clinical examination and medical imaging:
  * symptomatic CAM-FAI patients
  * asymptomatic CAM controls
  * healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Symptomatic CAM-FAI patients (Experimental): 33 patients that exhibit symptomatic CAM-FAI on medical imaging (Alpha angle >60) and have reduced hip internal rotation (IR<15). All participants in this group will be males aged between 21 and 35 years old.
  Interventions: Diagnostic Test: EOS; Diagnostic Test: 3D motion lab analysis
- Asymptomatic CAM-FAI patients (Experimental): 33 healthy control that exhibit asymptomatic CAM on x-ray scans (Alpha angle >60). All participants in this group will be males aged between 21 and 35 years old.
  Interventions: Diagnostic Test: EOS; Diagnostic Test: 3D motion lab analysis
- Healthy controls (Experimental): 33 healthy control that exhibit no symptoms or abnormal morphologies of the proximal femur (Alpha angle >60 , IR>15). All participants in this group will be males aged between 21 and 35 years old.
  Interventions: Diagnostic Test: EOS; Diagnostic Test: 3D motion lab analysis

INTERVENTIONS:
Diagnostic Test: EOS — Every subject in this study will undergo a radiographic analysis of the hip and spine using a low-dose, full-body biplanar X-ray acquisition (in standing, sitting and squatting position, EOS imaging).
Diagnostic Test: 3D motion lab analysis — A hip-specific 3D motion analysis will be performed. The 3D motion protocol will be divided into 2 main sections.
  First section: Consist of movements categorized within the activities of daily living (walking at self-selected speed, uphill walking, standardized deep squat and non-standardized deep squat)
  Second section: Consists of movements that are categorized within athletic training and have been specifically chosen to induce large hip ranges of motion (Sumo squats, dead lifts, forward lunges, running uphill and downhill)
  Each movements will be repeated 6 times. Three times with the dominant foot/opposite leg on the force plate to collect kinetic data. All data will be captured using two 10-15 camera 3D motion capture systems and one capturing an instrumented treadmill (M-gait)

SUMMARY:
Femoroacetabular impingement (FAI) is an orthopaedic condition that is primarily characterized by the presence of anatomic bony abnormalities in the femoral head and/or the acetabulum resulting in an abnormal contact between the two during hip motion, especially in positions of increased hip flexion and rotation, ultimately leading to hip pain. Unfortunately, a FAI diagnosis is frequently only made once symptoms have become severe to an extent that they limit everyday life activities. Moreover, another important aspect that has been consistently overlooked in past FAI movement studies is the influence muscle strength and activation can have on movement pattern and symptom presentation. The diagnosis and management of FAI needs to be addressed through a more wholesome investigation of the biomechanical influence on the manifestation of symptoms.

This project aims to further unravel the link between spinopelvic anatomy, its biomechanical contribution to femoro-pelvic motion and the manifestation of femoroacetabular impingement in adult male population. By, for the first time, integrating three-dimensional (3D) instrumented motion analysis with state-of-the-art full-body biplanar X-ray imaging (EOS imaging, Paris France), we will more specifically investigate the presence of an association between spinopelvic kinematics and the link to symptomatic FAI morphology, as well as investigate the presence of differences in these measures between symptomatic and asymptomatic subjects with comparable femoral morphology.

DETAILED DESCRIPTION:
Femoroacetabular impingement (FAI) is an orthopaedic condition that is primarily characterized by the presence of anatomic bony abnormalities in the femoral head and/or the acetabulum resulting in an abnormal contact between the two during hip motion, especially in positions of increased hip flexion and rotation, ultimately leading to hip pain. FAI can be radiologically classified into 3 types of morphology: Pincer, CAM and mixed type. While a clear-cut radiological classification makes the identification of FAI seem quite straightforward, it fails to differentiate between symptomatic and asymptomatic patients.

Unfortunately, a FAI diagnosis is frequently only made once symptoms have become severe to an extent that they limit everyday life activities. Not only this movement restriction is a significantly debilitating factor in such a young active population, a recent study reported FAI patients to see on average 4.0 health care providers, undergo on average 3.4 diagnostic imaging tests, and receive on average 3.1 treatments prior to final diagnosis. This raises the cost of an individual FAI diagnosis to be €1,563.26 higher than the calculated minimum required cost. Such calculations clearly reveal the long-lasting, multifactorial burden of FAI on society.

Moreover, another important aspect that has been consistently overlooked in past FAI movement studies is the influence muscle strength and activation can have on movement pattern and symptom presentation. To our knowledge only three studies have looked into muscle strength by using mainly hand-held dynamometers to record the isometric strength of hip musculature. Their findings suggest hip muscle weakness in symptomatic FAI subjects, but whether this weakness is a pain protective consequence, or an actual cause of FAI is still unknown.

In conclusion, the diagnosis and management of FAI needs to be addressed through a more wholesome investigation of the biomechanical influence on the manifestation of symptoms.

This project aims to further unravel the link between spinopelvic anatomy, its biomechanical contribution to femoro-pelvic motion and the manifestation of femoroacetabular impingement in adult male population. By, for the first time, integrating three-dimensional (3D) instrumented motion analysis with state-of-the-art full-body biplanar X-ray imaging (EOS imaging, Paris France), we will more specifically investigate the presence of an association between spinopelvic kinematics and the link to symptomatic FAI morphology, as well as investigate the presence of differences in these measures between symptomatic and asymptomatic subjects with comparable femoral morphology.

ELIGIBILITY:
Exclusion Criteria:

- Participants in all three study groups will be excluded if x-ray scans shows a pincer FAI morphology or radiological sign of osteoarthritis.

Inclusion Criteria:

* All participants will be males aged between 21 and 35 years old.
* For symptomatic CAM-FAI patients

  1. The presence of CAM-FAI morphology at the head-neck junction of the femur
  2. Alpha angle >60
  3. Reduced hip internal rotation (IR<15)
* For asymptomatic CAM controls:

  1. Exhibit asymptomatic CAM on x-ray scansAlpha angle >60
* For Healthy control group:

  1. Exhibit no symptoms or abnormal morphologies of the proximal femur (Alpha angle >60 , IR>15).

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The presence of CAM morphology in combination with symptoms | Baseline
  1. = yes morphology, yes symptoms;
  2. = yes morphology, no symptoms;
  3. = no morphology, no symptoms

SECONDARY OUTCOMES:
The Copenhagen Hip and Groin Outcome Score (HAGOS) | Baseline
  Consists of six separate subscales assessing Pain, Symptoms, Physical function in daily living, Physical function in Sport and Recreation, Participation in Physical Activities and hip and/or groin-related Quality of Life (QOL).
Radiographic spinopelvic parameters | Baseline
  Radiographic spinopelvic parameters will be collected via a radiographic analysis of the hip and spine using a low-dose, full-body biplanar X-ray acquisition (in standing, sitting and squatting position) as well as a classic x-ray image in 45° Dunn view of both hips.
3D motion analysis parameters | Baseline
  3D motion analysis parameters will be collected via a hipspecific 3D motion analysis where different movements will be performed on the force plate.

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Ghijselings, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals of Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No